CLINICAL TRIAL: NCT05471427
Title: Predictive fActors for toleraNce to Taxane Based CHemotherapy In Older adultS Affected by mEtastatic Prostate Cancer, a Prospective Observational Study (ANCHISES)
Brief Title: Predictive fActors for toleraNce to Taxane Based CHemotherapy In Older adultS Affected by mEtastatic Prostate Cancer
Acronym: ANCHISES
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: ANCHISES
Record Dates: First submitted 2022-07-08; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Elderly Patients; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; cabazitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Taxane chemotherapy — Patients underwent taxane chemotherapy according to clinical practice for metastatic prostate cancer
  Other Names: Docetaxel or Cabazitaxel

SUMMARY:
Aiming to explore predictive factors of fitness to taxane chemotherapy in elderly patients, the investigators collected data from a prospective mono-centric database of patients aged >/= 70 years old treated in our department, and explored association between baseline age, G8 score and Charlson comorbidity index with taxane dose reduction, treatment temporary suspension or definitive interruption.

DETAILED DESCRIPTION:
Patients included in the analysis were affected by metastatic prostate cancer with >/=70 years old. All patients underwent Taxane treatment starting with standard treatment schedules (75 mg/m2 or 25 mg/m2 every 3 weeks, respectively). Chemotherapy with Docetaxel was scheduled for a total of 6-8 cicles in the mHSPC-mCRPC setting, respectively, and up to 9 cycles for Cabazitaxel treatment.

Indication to taxane chemotherapy was based on treating physician choice. G8 Questionnaires were collected before start and at the end of chemotherapy. Charlson comorbidity index was recorded for all patients before chemotherapy start. Data comprehensive of age, castrate resistant status , type of taxane used , Growth factors use during treatment, previous and following treatment with ARTAs or other taxanes, number of cycles administered, dose reductions , treatment suspension and treatment definitive interruptions unrelated to progressive disease, were collected and reported. Logistic regression was performed to explore the association between outcomes and baseline age, CCI and G8 score. Receiver Operating Characteristic curves analysis was performed to look for the optimal cut-off value for features significantly associated with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by metastatic prostate cancer

  ->/=70 years old.
* Patients undergoing Taxane treatment with Docetaxel or Cabazitaxel

Exclusion criteria:

* Patients younger than 70 years old.
* Patients unsuitable for taxane chemotherapy

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients affected by metastatic prostate cancer (either in castrate resistant or hormone sensitive status), undergoing taxane chemotherapy in any setting at an age >/=70 years old
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment interruption | 10 months
  Number of participants with definitive treatment stop unrelated to treatment progression

SECONDARY OUTCOMES:
Treatment suspension | 10 months
  Number of participants with temporary treatment stop related to adverse event

OTHER OUTCOMES:
Dose reduction | 10 months
  Number of participants with dose schedule modification related to adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo LL Livi, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy

REFERENCES:
- [Background] Berthold DR, Pond GR, Soban F, de Wit R, Eisenberger M, Tannock IF. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer: updated survival in the TAX 327 study. J Clin Oncol. 2008 Jan 10;26(2):242-5. doi: 10.1200/JCO.2007.12.4008. PMID 18182665
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Kyriakopoulos CE, Chen YH, Carducci MA, Liu G, Jarrard DF, Hahn NM, Shevrin DH, Dreicer R, Hussain M, Eisenberger M, Kohli M, Plimack ER, Vogelzang NJ, Picus J, Cooney MM, Garcia JA, DiPaola RS, Sweeney CJ. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer: Long-Term Survival Analysis of the Randomized Phase III E3805 CHAARTED Trial. J Clin Oncol. 2018 Apr 10;36(11):1080-1087. doi: 10.1200/JCO.2017.75.3657. Epub 2018 Jan 31. PMID 29384722
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Gravis G, Fizazi K, Joly F, Oudard S, Priou F, Esterni B, Latorzeff I, Delva R, Krakowski I, Laguerre B, Rolland F, Theodore C, Deplanque G, Ferrero JM, Pouessel D, Mourey L, Beuzeboc P, Zanetta S, Habibian M, Berdah JF, Dauba J, Baciuchka M, Platini C, Linassier C, Labourey JL, Machiels JP, El Kouri C, Ravaud A, Suc E, Eymard JC, Hasbini A, Bousquet G, Soulie M. Androgen-deprivation therapy alone or with docetaxel in non-castrate metastatic prostate cancer (GETUG-AFU 15): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Feb;14(2):149-58. doi: 10.1016/S1470-2045(12)70560-0. Epub 2013 Jan 8. PMID 23306100
- [Background] Smith MR, Hussain M, Saad F, Fizazi K, Sternberg CN, Crawford ED, Kopyltsov E, Park CH, Alekseev B, Montesa-Pino A, Ye D, Parnis F, Cruz F, Tammela TLJ, Suzuki H, Utriainen T, Fu C, Uemura M, Mendez-Vidal MJ, Maughan BL, Joensuu H, Thiele S, Li R, Kuss I, Tombal B; ARASENS Trial Investigators. Darolutamide and Survival in Metastatic, Hormone-Sensitive Prostate Cancer. N Engl J Med. 2022 Mar 24;386(12):1132-1142. doi: 10.1056/NEJMoa2119115. Epub 2022 Feb 17. PMID 35179323
- [Background] Boyle HJ, Alibhai S, Decoster L, Efstathiou E, Fizazi K, Mottet N, Oudard S, Payne H, Prentice M, Puts M, Aapro M, Droz JP. Updated recommendations of the International Society of Geriatric Oncology on prostate cancer management in older patients. Eur J Cancer. 2019 Jul;116:116-136. doi: 10.1016/j.ejca.2019.04.031. Epub 2019 Jun 10. PMID 31195356
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Horgan AM, Seruga B, Pond GR, Alibhai SM, Amir E, De Wit R, Eisenberger MA, Tannock IF. Tolerability and efficacy of docetaxel in older men with metastatic castrate-resistant prostate cancer (mCRPC) in the TAX 327 trial. J Geriatr Oncol. 2014 Apr;5(2):119-26. doi: 10.1016/j.jgo.2013.12.001. Epub 2014 Jan 2. PMID 24495703
- [Background] Della Pepa C, Cavaliere C, Rossetti S, Di Napoli M, Cecere SC, Crispo A, De Sangro C, Rossi E, Turitto D, Germano D, Iovane G, Berretta M, D'Aniello C, Pisconti S, Maiorino L, Daniele B, Gridelli C, Pignata S, Facchini G. Predictive Comprehensive Geriatric Assessment in elderly prostate cancer patients: the prospective observational scoop trial results. Anticancer Drugs. 2017 Jan;28(1):104-109. doi: 10.1097/CAD.0000000000000428. PMID 27579728
- [Background] Gerritse FL, Meulenbeld HJ, Roodhart JM, van der Velden AM, Blaisse RJ, Smilde TJ, Erjavec Z, de Wit R, Los M; NePro Study Investigators. Analysis of docetaxel therapy in elderly (>/=70 years) castration resistant prostate cancer patients enrolled in the Netherlands Prostate Study. Eur J Cancer. 2013 Oct;49(15):3176-83. doi: 10.1016/j.ejca.2013.06.008. Epub 2013 Jul 9. PMID 23849828
- [Background] Maia MC, Pereira AAL, Lage LV, Fraile NM, Vaisberg VV, Kudo G, Barroso-Sousa R, Bastos DA, Dzik C. Efficacy and Safety of Docetaxel in Elderly Patients With Metastatic Castration-Resistant Prostate Cancer. J Glob Oncol. 2018 Sep;4:1-9. doi: 10.1200/JGO.2016.007807. Epub 2017 Mar 27. PMID 30241182
- [Background] Shayegan B, Wallis CJD, Hamilton RJ, Morgan SC, Cagiannos I, Basappa NS, Ferrario C, Gotto GT, Fernandes R, Roy S, Noonan KL, Niazi T, Hotte SJ, Saad F, Hew H, Park-Wyllie L, Chan KFY, Malone S. Real-world utilization and outcomes of docetaxel among older men with metastatic prostate cancer: a retrospective population-based cohort study in Canada. Prostate Cancer Prostatic Dis. 2023 Mar;26(1):74-79. doi: 10.1038/s41391-022-00514-9. Epub 2022 Feb 23. PMID 35197558
- [Background] Italiano A, Ortholan C, Oudard S, Pouessel D, Gravis G, Beuzeboc P, Bompas E, Flechon A, Joly F, Ferrero JM, Fizazi K. Docetaxel-based chemotherapy in elderly patients (age 75 and older) with castration-resistant prostate cancer. Eur Urol. 2009 Jun;55(6):1368-75. doi: 10.1016/j.eururo.2008.07.078. Epub 2008 Aug 8. PMID 18706755
- [Background] Takaha N, Okihara K, Kamoi K, Hongo F, Iwata T, Yano K, Ueda T, Takeuchi I, Yamada T, Kawauchi A, Miki T. Feasibility of tri-weekly docetaxel-based chemotherapy for elderly patients (age 75 and older) with castration-resistant prostate cancer. Urol Int. 2011;87(3):263-9. doi: 10.1159/000328217. Epub 2011 Aug 26. PMID 21876321
- [Background] Wang KY, Ma L, Zhang LL, Hu YC, Jiang JH, Ma Q. Efficacy and safety of docetaxel and prednisolone chemotherapy in very elderly men with metastatic castration-resistant prostate cancer (mCRPC) in real world: a single institute experience. Ann Palliat Med. 2021 Feb;10(2):1438-1444. doi: 10.21037/apm-20-573a. Epub 2020 Oct 15. PMID 33081478
- [Background] Kellokumpu-Lehtinen PL, Harmenberg U, Joensuu T, McDermott R, Hervonen P, Ginman C, Luukkaa M, Nyandoto P, Hemminki A, Nilsson S, McCaffrey J, Asola R, Turpeenniemi-Hujanen T, Laestadius F, Tasmuth T, Sandberg K, Keane M, Lehtinen I, Luukkaala T, Joensuu H; PROSTY study group. 2-Weekly versus 3-weekly docetaxel to treat castration-resistant advanced prostate cancer: a randomised, phase 3 trial. Lancet Oncol. 2013 Feb;14(2):117-24. doi: 10.1016/S1470-2045(12)70537-5. Epub 2013 Jan 4. PMID 23294853
- [Background] Sternberg CN, Castellano D, de Bono J, Fizazi K, Tombal B, Wulfing C, Kramer G, Eymard JC, Bamias A, Carles J, Iacovelli R, Melichar B, Sverrisdottir A, Theodore C, Feyerabend S, Helissey C, Poole EM, Ozatilgan A, Geffriaud-Ricouard C, de Wit R. Efficacy and Safety of Cabazitaxel Versus Abiraterone or Enzalutamide in Older Patients with Metastatic Castration-resistant Prostate Cancer in the CARD Study. Eur Urol. 2021 Oct;80(4):497-506. doi: 10.1016/j.eururo.2021.06.021. Epub 2021 Jul 15. PMID 34274136